CLINICAL TRIAL: NCT05192590
Title: Establishing Clinical Utility Evidence for Chronic Disease Management Testing (CDMT): A CPV® RandomizedControlled Trial
Brief Title: Establishing Clinical Utility Evidence for Chronic Disease Management Testing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Qure Healthcare, LLC (Industry)
Responsible Party: Principal Investigator, David Paculdo, Principle Investigator, Qure Healthcare, LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00057790
Record Dates: First submitted 2021-10-27; First posted 2022-01-14 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Cardiometabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: The study will enroll primary care physicians practicing in the US. Participants are randomly assigned to either control, intervention 1, or intervention 2 arms upon enrollment. All eligible and consented participants will complete two rounds of three patient simulations.
  The intervention 1 and intervention 2 arms only will receive educational material about the Aegis test in between these two rounds. Intervention 1 arm participants only will receive the CDMT results whether they select it or not, and Intervention 2 participants will receive the CDMT results only if they select it in the second round of simulated cases
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): These providers will complete two rounds of three simulated patient cases (CPVs). Control arm physicians will continue to have access to standard of care diagnostic tools, but not the CDMT test results.
- Educational Materials and CDMT Test Results (Intervention 1) (Experimental): Participants will care for the same set of CPV patients as the control arm, but will be educated on and will receive the CDMT test results whether they select it or not. Investigators will compare intervention participants' clinical recommendations to those in the control arm.
  Interventions: Other: Educational Materials and Chronic Disease Management Test (CDMT)
- Educational Materials and CDMT Test Results when Selected (Intervention 2) (Experimental): Participants will care for the same set of CPV patients as the control arm, but will be educated on and will receive the CDMT test results only if they select it. Investigators will compare intervention participants' clinical recommendations to those in the control arm.
  Interventions: Other: Educational Materials and Chronic Disease Management Test (CDMT)

INTERVENTIONS:
Other: Educational Materials and Chronic Disease Management Test (CDMT) — Intervention-1- and Intervention-2-arm participants will receive educational materials duplicating what physicians would receive in the real-world market as they adopt the CDMT technology. These materials are comprised of a PowerPoint presentation.
  Intervention 1 participants only will receive the CDMT test results whether they select it or not, and Intervention 2 participants will receive the CDMT test results only if they select it during the second round of case simulations.
  Arms: Educational Materials and CDMT Test Results (Intervention 1); Educational Materials and CDMT Test Results when Selected (Intervention 2)

SUMMARY:
This is a national-level research study of primary care physicians. The purpose of this study is to assess the clinical evaluation and management (drug, procedures, counseling and other) of a subset of common patient care indications.

DETAILED DESCRIPTION:
The results of this study could contribute to improved quality of care for patients by encouraging better care practices and adherence to evidence-based guidance. The data from this study will be submitted to a national journal for publication. The study plans to enroll up to 300 physicians.

Upon consenting and agreeing to participate in this study, participants will be asked to care for 3 simulated patient cases, known as Clinical Performance and Value Vignettes (CPV®). CPVs describe patients physicians typically encounter in their daily practice and are not meant to be difficult. In each vignette, physicians are asked to share their expected care through 5 domains: 1) history, 2) physical exam, 3) diagnostic workup, 4) diagnosis and 5) treatment and follow-up. Each case takes approximately 15-20 minutes to complete and we estimate the time commitment for each round of CPV administration to be approximately 45 - 60 minutes. All responses to the cases will be completed online and will be kept confidential. Over 2 CPV administration rounds, the total time to care for the simulated patients is estimated at 1.5-2 hours.

If physicians are randomized to an intervention group in this study, they will receive education materials on a diagnostic test currently available for use in the market after the first round of CPV administration. They are asked to review these materials before moving to the next CPV administration round. Time to review education materials is estimated to be approximately 15 minutes.

Depending on the results of this randomized controlled trial, there may be an opportunity for physicians to re-enroll into a follow-on study. If they choose to participate in this second study, they will be asked to identify and send de-identified records of patients in their practice that are similar to the simulated patients they previously cared for in this study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet the following criteria to be enrolled in the study:

  1. Board-certified physician currently practicing in the following areas:

     1. Internal medicine
     2. Family medicine
  2. Have practiced as a board-certified physician in internal or family medicine or greater than 2 but less than 30 years
  3. Community / non-academic based practice setting
  4. ≥ 40 patients under care weekly
  5. Commonly treats patients with atrial fibrillation, coronary artery disease, congestive heart failure, diabetes, hypertension, and hyperlipidemia
  6. Practicing in the U.S.
  7. English-speaking
  8. Access to the internet
  9. Informed and voluntarily consented to be in the study

Exclusion Criteria:

1. Non-English speaking
2. Practicing in an academic setting
3. Unable to access the internet
4. Not practicing in the U.S.
5. Do not voluntarily consent to be in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 249 (Estimated)
Dates: Start 2021-10-22 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2023-02-22 (Estimated)

PRIMARY OUTCOMES:
CPV-measured clinical score difference(drug, procedures, counseling and other) | 12 months
  Difference-in-differences regression analysis between the control and the intervention groups' diagnosis and treatment of chronic dyspnea, as measured by the participants diagnostic and treatment CPV case domain scores. In each domain of a CPV (history, physical exam, workup, diagnosis and treatment), participants' care recommendations are evaluated against evidence-based care scoring criteria which can sum from 0 to a high potential score of up to 100 percent in each domain, where higher scores mean better outcomes.
Test Adoption Rate | 12 months
  Rate of adoption of the CDMT test in Intervention 2 arm participants.
CPV-measured cost difference | 12 months
  Difference in expected cost of care between control and intervention participants. (Cost will be calculated by measuring differential rates of medical interventions/levels of care selected by each arm, and multiplying by Medicare reimbursement rates for these interventions, and/or by modeling the incidence of expected complications and calculating associated costs.)

SECONDARY OUTCOMES:
CPV-measured clinical score differences by use case | 12 months
  Difference in the overall, and the diagnostic and treatment quality scores between control and intervention participants. Diagnostic and treatment scores are calculated as the percent correct on CPVs, and the overall score is a average score of the subcategory scores (percent correct). This will be examined for each of the use cases to determine in which case(s) CPV scores most improved.
CPV-measured cost differences by use case | 12 months
  Difference in expected cost of care between control and intervention participants. (Cost will be calculated by measuring differential rates of medical interventions/levels of care selected by each arm, and multiplying by Medicare reimbursement rates for these interventions, and/or by modeling the incidence of expected complications and calculating associated costs.) This will be examined for each of the use cases to determine in which case(s) cost metrics most improved.
CPV-measured baseline variation | 12 months
  Participants completing the simulated cases, or CPVs, receive scores based upon the quality of care they provide. This measure will assess the baseline levels of variation in the care of pain patients among all participants, including by use case types

CONTACTS AND LOCATIONS:
Locations (1):
- QURE Healthcare, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peabody JW, Ganesan D, Valdenor C, Paculdo D, Schrecker J, Westerfield C, Heltsley R. Randomized prospective trial to detect and distinguish between medication nonadherence, drug-drug interactions, and disease progression in chronic cardiometabolic disease. BMC Prim Care. 2023 Apr 15;24(1):100. doi: 10.1186/s12875-023-02042-4. PMID 37061690
- [Derived] Valdenor C, Ganesan D, Paculdo D, Schrecker J, Heltsley R, Westerfield C, Peabody JW. Clinical Variation in the Treatment Practices for Medication Nonadherence, Drug-Drug Interactions, and Recognition of Disease Progression in Patients with Chronic Cardiometabolic Diseases: A Cross-Sectional Patient Simulation Study among Primary Care Physicians. Int J Clin Pract. 2022 Jul 30;2022:6450641. doi: 10.1155/2022/6450641. eCollection 2022. PMID 35989865